CLINICAL TRIAL: NCT00824824
Title: Effect of Cosopt Versus Combigan on Retinal Vascular Autoregulation in Primary Open Angle Glaucoma (POAG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Louis Pasquale, MD, Director, Glaucoma Service Associate Director, Telemedicine, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 08-12-057
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Results first posted 2016-10-28 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Glaucoma
Keywords: Retinal Vascular Autoregulation
MeSH Terms: conditions — Glaucoma | interventions — dorzolamide; dorzolamide-timolol combination; Brimonidine Tartrate; Brimonidine Tartrate, Timolol Maleate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brimonidine 0.2%-timolol 0.5% arm (Experimental): Patients using timolol were switched to brimonidine tartrate / timolol maleate 0.2%/05% 1 get BID OU for six weeks.
  Interventions: Drug: Brimonidine 0.2%-0.5% timolol 0.5
- Dorzolamide 2%-timolol 0.5% arm (Active Comparator): Patients using timolol were switched ti dorzolamide hydrochloride / timolol 0.5% 2%/0.5% bid OU for six weeks
  Interventions: Drug: Dorzolamide 2%-timolol 0.5%

INTERVENTIONS:
Drug: Dorzolamide 2%-timolol 0.5% — BID OU for 6 weeks
  Other Names: Cosopt; RVD intervention after run-in on timolol 0.5% bid OU
  Arms: Dorzolamide 2%-timolol 0.5% arm
Drug: Brimonidine 0.2%-0.5% timolol 0.5 — BID OU for 6 weeks
  Other Names: Combigan; RVD intervention after run-in on timolol 0.5% bid OU
  Arms: Brimonidine 0.2%-timolol 0.5% arm

SUMMARY:
We have completed a study in which we examined the response of the retinal circulation to changes in posture from sitting to lying down in patients with primary open angle glaucoma (POAG). This alteration in position produces changes in the local blood pressure at the entrance to the retinal vasculature. In a healthy retina, the vasculature adapts by dilating and constricting in order to maintain a steady blood flow rate. In an eye with POAG, this often does not occur. As a result, there are large fluctuations in blood flow which may produce the retinal neuronal damage associated with glaucoma.

The purpose of this study is to demonstrate that topical anti-glaucoma treatments with agents that have vasoactive as well as IOP-lowering effects can have a beneficial effect on maintaining a steady retinal blood flow rate even when there are changes in local blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* POAG
* Age 40 to 80 years
* Untreated IOP greater than 21 mm Hg

Exclusion Criteria:

* More than two IOP lowering medications
* Exfoliation or pigment dispersion syndrome
* Diabetic retinopathy
* History of ocular surgery

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis Pasquale, Principal Investigator — Mass Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feke GT, Pasquale LR. Retinal blood flow response to posture change in glaucoma patients compared with healthy subjects. Ophthalmology. 2008 Feb;115(2):246-52. doi: 10.1016/j.ophtha.2007.04.055. Epub 2007 Aug 8. PMID 17689612

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 21 primary open angle glaucoma patients were recruited for the study from the practices of Douglas J. Rhee, Angela V. Turalba, and Louis R. Pasquale at Massachusetts Eye and Ear Infirmary, Boston. Recruitment took place between February 13, 2009 and December 21, 2011.
Pre-assignment Details: Prior to the initial testing visit, subjects ceased using their current IOP-lowering medications and were run in for 6 weeks on timolol 0.5% BID OU. After this 6 week period baseline measurements were taken and 7 were identified with retinal vascular dysregulation. These 7 patients were then randomized into one of two treatment arms.
Groups:
- Dorzolamide-Timolol Then Brimonidine-Timolol: 4 of the 7 POAG subjects with RVD were randomized into the dorzolamide hydrochloride 2% - timolol 0.5% ophthalmic solution. The 4 subjects received this treatment for 6 weeks. After the 6-week period the same measurements that were taken at baseline where taken once again. After these measurements were collected these 4 subjects were treated with brimonidine tartrate 0.2%-timolol maleate 0.5% ophthalmic solution for 6 weeks. After this second 6 week period the same measurements that were taken previously were taken again.
- Brimonidine-Timolol Then Dorzolamide-Timolol: 3 of the 7 POAG RVD subjects were ransomized into the brimonidine tartrate 0.2%-timolol maleate 0.5% ophthalmic solution. The 3 subjects received this treatment for 6 weeks. After the 6-week period the same measurements that were taken at baseline where taken once again. After these measurements were collected these 3 subjects were treated with dorzolamide hydrochloride 2% - timolol 0.5% ophthalmic solution for 6 weeks.After this second 6 week treatment period the same measurements where taken again.
Period: Overall Study
Arm/Group | Dorzolamide-Timolol Then Brimonidine-Timolol | Brimonidine-Timolol Then Dorzolamide-Timolol
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There are 14 subjects in this study whop have PAOG without RVD. There are 7 subjects with POAG with RVD. The 14 subjects without RVD did not continue in the two treament arms of this study.
Groups:
- Primary Open Angle Glaucoma: Subjects of either gender with age range 40 to 80 years old with POAG were eligible for the study. Eligible subjects had a history of an untreated IOP > 21 mmHg in the left eye and a CPSD ≥ 1.0 in this eye. Patients being treated with more than two IOP lowering medications concurrently were excluded. All eligible subjects had open angles on gonioscopy with the filtering portion of the trabecular meshwork visible for 360° in both eyes. All subjects also had at least two reliable Humphrey 24-2 full threshold visual fields that showed reproducible loss in the left eye on tests with fixation loss ≤33%, false positives ≤ 20% and false negatives ≤ 20%. Patients with evidence of exfoliation or pigment dispersion syndrome in either eye were excluded. Subjects with diabetic retinopathy or a history of ocular laser or incisional surgery in either eye were also excluded.
- POAG With RVD: 7 subjects with POAG were identified to have retinal vascular dysregulation (RVD). We determined whether RVD was present in the following way. The percentage change between the retinal blood flow measured while reclining for 30 min and the baseline retinal blood flow measured while seated was calculated. In a previous study, we found that among healthy subjects the change in the retinal blood flow while reclining compared to sitting was +6.5% ± 12%. For this study, we defined the normal range of blood flow autoregulation as ±2 standard deviations about the mean percentage change found in the control group in our previous study. Subjects with a change in retinal blood flow induced by posture change outside of -17.5% to +35.5% where considered to have RVD.
- Total: Total of all reporting groups
Arm/Group | Primary Open Angle Glaucoma | POAG With RVD | Total
Number analyzed (Participants) | 14 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (8.2) | 60.0 (8.6) | 63 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 11 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 13 | 7 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Presence of Retinal Vascular Dysregulation (RVD)
Description: We determined whether RVD was present in the following way. The difference between the retinal blood flow measured while reclining for 30 minutes and the baseline retinal blood flow measured while seated was calculated. In a previous study, we found that among healthy subjects the change in the blood flow while reclining compared to baseline was +6.5% ± 12%. For this study, we defined the normal range of blood flow autoregulation as ± 2 standard deviations about the mean percentage change found in the control group in the initial study (6.5% ± 24.0%); that is, as -17.5% to +30.5%. Participants with a change in retinal blood flow induced by posture change outside this range were randomized to either dorzolamide-timolol fixed combination BID OU or brimonidine-timolol fixed combination BID OU for 6 weeks.
Time Frame: 6 weeks post treatment
Population: 21 participants were tested for RVD after 6 weeks of timolol treatment. Of the 21 participants who were tested, 7 had RVD and were randomized to Dorzolamide-Timolol and Brimonidine-Timolol; 14 had normal autoregulation. One participant was removed from the analysis in the Brimonidine-Timolol arm due to technical difficulties with equipment.
Measure: Number; unit: Participants
Groups:
- Dorzolamide-Timolol: Post timolol-dorzolamide outcome: All 7 patients who had RVD following timolol had retinal vascular autoregulation that was in the normal range.
- Brimonidine-Timolol: Post timolol-brimonidine outcome: 6 of the 7 patients were tested following timolol-brimonidine. One of the 7 patients could not be tested due to technical issues. Of the 6 that were tested, 4 patients had retinal vascular autoregulation that was in the normal range. Two patients continued to show RVD.
Arm/Group | Dorzolamide-Timolol | Brimonidine-Timolol
Number analyzed (Participants) | 7 | 6
Participants | 7 | 4

ADVERSE EVENTS:
Time Frame: The time period of the entire study.
Arm/Group | Dorzolamide-Timolol Then Brimonidine-Timolol | Brimonidine-Timolol Then Dorzolamide-Timolol
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

LIMITATIONS AND CAVEATS:
A potential limitation of this study is that no washout period occurred because the 6-week treatment periods extended beyond the typical 2-week washout period for dorzolamide and the 3-week washout period for brimonidine.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No